CLINICAL TRIAL: NCT03978325
Title: Preoperative Exercise to Improve Fitness in Patients Undergoing Complex Surgery for Cancer of the Lung or Oesophagus
Brief Title: Preoperative Exercise for Patients Undergoing Complex Cancer Surgery
Acronym: PRE-HIIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Health Research Board, Ireland (Other); Irish Cancer Society (Other)
Responsible Party: Principal Investigator, Prof Juliette Hussey, Professor of Physiotherapy, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pre-HIIT
Record Dates: First submitted 2019-05-17; First posted 2019-06-07 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Complications; Physical Activity; Surgery--Complications
Keywords: Prehabilitation; Exercise; Surgery
MeSH Terms: conditions — Postoperative Complications; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): This arm will complete a standard prehabilitation intervention.
  Interventions: Other: Control
- HIIT Intervention (Experimental): This group will complete a pre-operative high intensity interval training programme.
  Interventions: Other: Exercise - HIIT Intervention

INTERVENTIONS:
Other: Control — The control group will receive standard pre-operative care. This involves standard pre-operative advice and a moderate intensity preoperative exercise programme.
  Arms: Control
Other: Exercise - HIIT Intervention — The HIIT intervention will take the form of a supervised programme, completed for at least two weeks, up to 5 days per week preoperatively. The HIIT intervention will be performed on a cycle ergometer. Exercise sessions will be individually supervised and scheduled at a time of convenience for each participant. Each exercise session will last 40 minutes and will include warm-up, exercise training and cool-down components. Lactate threshold, measured during the baseline CPT, will be used to determine the exercise intensity.
  The training protocol will prescribe 15 second intervals of exercise and passive recovery. The highest resistance reached during the baseline CPET (measured in watts) will be recorded as the peak power output (PPO). During training, participants will undergo a 5-minute warm-up at 50% PPO, followed by up to 30 minutes of HIIT with intervals of 15 seconds at 100% PPO with 15 second recovery periods at 0 watts.
  Arms: HIIT Intervention

SUMMARY:
Treatment for people with cancer of the lung or the oesophagus (food-pipe) often involves surgery. This surgery is complex and there is a high risk that patients will develop severe complications afterwards, leading to a longer hospital stay and higher hospital costs, and impacting greatly on recovery and quality of life. If patients' lungs and heart can be optimised before surgery, then recovery may be improved. While fitness can be improved by exercise, the lead-in time to surgery following a cancer diagnosis is often very short, and research is needed to examine what types of exercise might be most effective at increasing fitness over a short period.

This project will investigate if high intensity interval training (HIIT) can increase fitness levels in people scheduled for surgery for cancer of the oesophagus or the lungs. HIIT alternates between periods of high intensity exercise, cycling on a stationary bike, followed by a period of more relaxed exercise. This approach is known to improve fitness but has not previously been investigated in patients awaiting complex cancer surgery.

Groups will be compared for changes in pre-surgery fitness levels, any complications they may experience after surgery, general physical recovery after surgery and the cost of care after surgery. The investigators anticipate that patients who undergo HIIT before surgery will have less complications and better recovery after surgery, a significantly improved quality of life, and lower costs of care.

DETAILED DESCRIPTION:
Patients with cancer of the lung or oesophagus, undergoing curative treatment, usually require a thoracotomy and a complex oncological resection. These surgeries carry a risk of major morbidity and mortality, and risk assessment, preoperative optimisation, and enhanced recovery after surgery (ERAS) pathways are modern approaches to optimise outcomes. Pre-operative fitness is an established predictor of postoperative outcome, accordingly targeting pre-operative fitness through exercise prehabilitation has logical appeal. Exercise prehabilitation is challenging to implement however due to the short opportunity for intervention between diagnosis and surgery. Therefore, individually prescribed, intensive exercise training protocols which convey clinically meaningful improvements in cardiopulmonary fitness over a short period need to be investigated. This project will examine the influence of exercise prehabilitation on physiological outcomes and postoperative recovery, evaluation of health economics, the impact of the programme on hospital costs.

This study will take the form of a randomised controlled trial aimed primarily at improving pre-operative fitness with high intensity interval training (HIIT). HIIT prescribes aerobic exercise which alternates between periods of high intensity training and active recovery. This form of exercise training stimulates greater improvements in cardiopulmonary fitness over short periods compared to continuous aerobic training and therefore may be ideally suited to exercise prehabilitation. The primary outcome, cardiopulmonary fitness, will be measured by cardiopulmonary exercise testing and explored further using a suite of pulmonary and physical performance measures. Secondary outcomes will examine the impact of individually prescribed HIIT on postoperative outcome, postoperative physical recovery, restoration of pre-treatment fitness levels and both acute and sub-acute hospital costs. The investigators anticipate that this mode of exercise prehabilitation will attenuate postoperative risk and improve postoperative recovery, thus improving patient quality of life and having considerable economic benefits for the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for either oesophagectomy (2-stage or 3-stage) or major lung resection for the management of primary oesophageal or lung cancer.
* Date of surgery ≥ 2 weeks from baseline assessment
* Ability to provide written informed consent
* Absence of significant co-morbidities, including metastatic disease, which may adversely impact postoperative outcome
* Successful completion of a medically supervised cardiopulmonary exercise test
* Patients with oesophageal cancer scheduled for multimodal therapy including preoperative chemo(radio)therapy and oesophagectomy will be recruited and tested prior to treatment commencement.

Exclusion Criteria:

* The American Thoracic Society/American College of Chest Physicians (ATS/ACCP) absolute contraindications for exercise testing will be applied.
* Patients undergoing video assisted lobectomy for early lung cancer will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1)
  Cardiorespiratory fitness will be determined by Cardiopulmonary Exercise Test (CPET)

SECONDARY OUTCOMES:
Clavien-Dindo Scale | At hospital discharge (approximately 7-14 days postoperatively)
  Measurement of the most severe complication that occurs in the postoperative period. The ordinal scale is divided into seven grades (Grade I-V, two sub-groups each for Grade III and IV), ranging from Grade I, which considers any deviation from normal, to Grade V, which describes death of the patient.
Change in the Post-Operative Morbidity Score (POMS) | On postoperative day 5, postoperative day 7 and at hospital discharge (approximately 7-14 days postoperatively)
  The POMS is a nine-domain tool that prospectively describes and records in-hospital postoperative complications following major surgery.
The Comprehensive Classification Index (CCI) | At hospital discharge (approximately 7-14 days postoperatively)
  This is a summary of overall morbidity including the type, number and severity of each complication experienced during the postoperative period.
Change in Pulmonary function | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1)
  Pulmonary function will be measured as the first step of the CPET. This will be used to determine forced vital capacity (FVC), forced expiratory volume at 1s (FEV1) and the ratio of FEV1/FVC.
Change in Maximum Inspiratory pressure | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1)
  PImax will measured using a PowerBreathe K-series portable respiratory pressure metre. Patients will be measured at residual volume during a forceful inspiratory manoeuvre while resting in a seated position.
Change in Muscle strength | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1)
  Quadriceps muscle strength will be measured by 1 repetition maximum (1RM) in kg's using a horizontal leg extension. The 1RM is defined as the highest load that can be lifted through full range of movement at one time.
Change in Self reported physical activity: International Physical Activity Questionnaire (IPAQ) | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1) as well as post-operative day 30
  This questionnaire evaluates activity in metabolic equivalent (MET)-hours per week over the previous seven days. The questionnaire also quantifies average weekend and weekday sitting time. The questionnaire also quantifies average weekend and weekday sitting time.
Change in Self reported functional recovery | At post-operative day 30
  Participants will rate their recovery as 0%, 25%, 50%, 75% or 100% according to standardised descriptors.
Change in Functional Performance | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1)
  This will be measured using the Short Physical Performance Battery (SPPB). This measure combines the results of gait speed, chair stand and balance tests. A score lower than 10 indicates one or more mobility limitations.
Change in Quality of Life | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1) and on post-operative day 30.
  Quality of Life will be determined by the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30).
  Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Change in Quality of Life (Specific to Lung Cancer) | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1) and on post-operative day 30.
  For Oesophago-gastric Cancer Patients Quality of Life will be further assessed with the European Organisation for Research and Treatment of Cancer Oesophago-gastric Cancer Subscale the EORTC QLQ-LC 13. Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Change in Quality of Life (Specific to Oesophageal Cancer) | At diagnosis (Dx), baseline (T0), immediately post-intervention (T1) and on post-operative day 30.
  For Oesophago-gastric Cancer Patients Quality of Life will be further assessed with the European Organisation for Research and Treatment of Cancer Oesophago-gastric Cancer Subscales the EORTC QLQ-OES18 and QLQ-OES25. Scores are reported on a linear scale from 0-100. A high score in a functional scale indicates greater function. A high score in a symptom scale indicates greater symptom burden.
Cost Effectiveness | At routine post-operative clinic visits at 6 weeks and 3 months postoperatively.
  The costs of the program will be set against the effects on HRQOL
Qualitative Approach | Immediately after the programme intervention (T1)
  Focus groups and interviews will be carried out with participants to gain their perspectives of the impact of the program on physical and mental well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Hussey, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- University of Dublin, Trinity College, Dublin, Ireland

REFERENCES:
- [Derived] Sheill G, Guinan E, O'Neill L, Normand C, Doyle SL, Moore S, Newell J, McDermott G, Ryan R, Reynolds JV, Hussey J. Preoperative exercise to improve fitness in patients undergoing complex surgery for cancer of the lung or oesophagus (PRE-HIIT): protocol for a randomized controlled trial. BMC Cancer. 2020 Apr 15;20(1):321. doi: 10.1186/s12885-020-06795-4. PMID 32293334